CLINICAL TRIAL: NCT00004324
Title: Developmental Phenomenology of Obsessive Compulsive Disorder and Tourette Syndrome in Children and Adolescents
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Yale University (Other)
Other Study IDs: NCRR-M01RR06022-5099; YALESM-5099
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-01

CONDITIONS: Tourette Syndrome; Obsessive Compulsive Disorder
Keywords: Tourette syndrome; anxiety disorder; disease-related problem/condition; neurologic and psychiatric disorders; obsessive compulsive disorder; oncologic disorders; rare disease
MeSH Terms: conditions — Tourette Syndrome; Obsessive-Compulsive Disorder; Anxiety Disorders; Neurologic Manifestations; Mental Disorders; Rare Diseases

SUMMARY:
OBJECTIVES: I. Characterize the natural history, associated features, and severity of symptoms of obsessive compulsive disorder and Tourette syndrome in children and adolescents.

II. Identify factors that influence the clinical course and prognosis of these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: All patients and their families participate in 6 parts of the study: current severity of symptoms, coincident disease diagnoses, natural history, neuropsychologic assessment, physical and neurologic assessment, and family history and function. The evaluations include the following: Current Severity of Symptoms Assessment, Children's Yale Brown Obsessive Compulsive Scale (CY-BOCS), Clinician's Global Impression-Obsessive Compulsive Disorder (CGI-OC), Leyton Obsessional Inventory-Child Version (LOI-CV), Obsessive Compulsive Personality Rating Scale, Yale Global Tic Severity Scale(YGTSS), Clinician's Global Impression-Tourette Syndrome (CGI-TS), Tourette Syndrome Symptom List (TSSL), Clinician's Global Impression-Anxiety (CGI-A), Covi Anxiety Scale (CAS), Children's Manifest Anxiety Scale-Revised (CMAS-R), Social Anxiety Scale for Children-Revised, Fear Survey Schedule for Children-Revised, Louisville Fear Survey, Children's Depression Rating Scale-Revised (CDRS-R), Clinician's Global Impression-Depression (CGI-D), Children's Depression Inventory (CDI), The Dimensions of Temperament Survey (DOTS), Mosher Guilt Scale-Revised, Real vs. Ideal Self Questionnaire, Harter Self-Perception Profile For Children, The Children's Global Assessment Scale (CGAS), The Child Behavior Checklist (CBCL), Coincident Disease Diagnoses Assessment, Diagnostic Interview Schedule for Children-II (DISC-II), Yale Best Estimate of Diagnoses Schedule (Y-BEDS), Natural History Evaluation, Yale Natural History Questionnaire (YHNQ), Social Readjustment Scale for Children, Neuropsychologic Assessment, Delayed Response Tasks, Continuous Performance Task, Continuous Recognition Memory, Selective Reminding Procedures, Card Sorting Tasks, Wechsler Intelligence Scale for Children-Revised, Digit Span, Digit Symbol and Mazes Paced Auditory, Serial Addition Task, Purdue Pegboard Trail Making Tasks, Fluency Tasks, Rey-Osterreith Complex Figure Stanford-Binet Intelligence Scale-Fourth Edition, Physical, Neurologic, and Neurochemical Assessment Physical exam (abbreviated), Physical and Neurological Examination for Soft Signs (PANESS), 24-hour urinary cortisol and catecholamines, Family History and Family Function Assessment of family history, Assessment of Family Functioning.

The estimated duration of study is 10 years.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Obsessive compulsive disorder or Tourette syndrome meeting Diagnostic and Statistical Manual of Mental Disorders IV criteria

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90
Dates: Start 1989-12

CONTACTS AND LOCATIONS:
Overall Officials: James F. Leckman, Study Chair — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States